CLINICAL TRIAL: NCT05815030
Title: PrEP4Kink: Testing the Effects of an Interactive Educational Intervention on PrEP Uptake Among Kink-Involved Adults
Brief Title: HIV Pre-Exposure Prophylaxis Among an Unrecognized Sexual Minority Population
Acronym: PrEP4Kink
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty enrolling participants in study created too long a delay
Sponsor: The Alternative Sexualities Health Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: T2022-02
Record Dates: First submitted 2022-11-16; First posted 2023-04-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: PrEP; HIV Prevention; Kink

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): experimental group, receiving 3 exposures to the kink-focused video intervention
  Interventions: Other: video informational/educational intervention
- Group B (Other): control group, receiving no exposure to the kink-focused video, but seeing the generic / standard video
  Interventions: Other: video informational/educational intervention
- Group C (Other): group that receives 1 exposure to the generic / standard video, and later 2 exposures to the kink-focused video
  Interventions: Other: video informational/educational intervention
- Group D (Other): group that receives 2 exposures to the generic / standard video, and later 1 exposure to the kink-focused video
  Interventions: Other: video informational/educational intervention

INTERVENTIONS:
Other: video informational/educational intervention — Videos relating to PrEP use, its benefits, side effects, and other information. The educational/round-table video will highlight individuals from diverse backgrounds and identities who will share their experiences using PrEP, including perceived benefits and effectiveness, experienced barriers to PrEP uptake, their reasons for using PrEP, and their own self-efficacy. The control group's (generic / standard video) materials will be focused on PrEP uptake without a kink identity perspective. The treatment group's materials, however, will include videos that feature kink-identified individuals who discuss PrEP uptake through a kink perspective.

SUMMARY:
The Alternative Sexualities Health Research Alliance (TASHRA) will work collaboratively with Gilead Sciences, Inc. to study Pre-Exposure Prophylaxis (PrEP) uptake and adherence; levels of stigma around PrEP use; and changes in health beliefs around PrEP use. The study design will compare kink-involved or bondage/discipline/dominance/submission/sadism/masochism (BDSM)-involved individuals responses to generic vs. kink-focused printed and educational-entertaining video materials in a 12 month crossover study.

The primary objective of the study is to examine factors that increase the uptake of PrEP in a novel sexual subculture by testing the impact of an entertainment-education intervention designed to be highly relatable to kink-involved individuals.

Secondary Objectives: PrEP4Kink will measure knowledge of PrEP and attitudes towards PrEP uptake over time. These are elements identified by the Health Belief Model: perceived risk of HIV; susceptibility to HIV; perceived barriers to PrEP uptake; perceived benefits of PrEP uptake; perceived effectiveness of PrEP; and self-efficacy of initiating PrEP uptake. Moderating and ancillary factors will be measured, and their relation to the elements of the Health Belief Model will be analyzed. Moderating factors include the centrality of kink identity; the level of kink community involvement; the types and frequencies of kink and sex behaviors. Demographic variables will be measured and their relation to elements of the Health Belief Model will be analyzed, including age; number of years involved in kink; gender identity; sex assigned at birth; racial/ethnic identity; educational attainment; income level; insurance coverage; sexual orientation identity; and sexual attraction.

DETAILED DESCRIPTION:
The primary objective of the study is to examine factors that increase the uptake of PrEP in a novel sexual subculture by testing the impact of an entertainment-education intervention designed to be highly relatable to kink-involved individuals.

In TASHRA's 2016 Kink Health Survey of 1,139 kink-involved individuals, the rate of HIV was approximately 10 times the national index. 37 (80.4%) of a total of 46 persons living with HIV were cis-male men who have sex with men (MSM) and men who have sex with men and women (MSMW). Seven (15.2%) were persons who had ever used intravenous drugs. Of those living with HIV, 38 (82.6%) were engaged in kink activities at high risk of blood exposure, 8 (17.4%) were engaged in activities at low risk of blood exposure, and none were engaged only in activities considered to have no risk of blood exposure. It should be noted that the sample for the 2016 Kink Health Survey was limited in racial and ethnic diversity, while having a high degree of gender and sexual orientation diversity.

Educational interventions appear to be effective in increasing PrEP uptake. One study of 116 African American women found that an avatar-led eHealth video that focused on education about PrEP from relatable characters did have a significant impact on intentions to seek out PrEP and to recommend PrEP to other women. Social cognitive theory predicts that perceived similarity of models enhances imitation and observational learning (together called vicarious learning). Social cognitive theory also proposes efficacy as an important element in the learning process by enhancing perseverance in learning and behavior. Efficacy is strongly affected by vicarious learning opportunities and verbal persuasion, which are key pathways for entertainment-education interventions. Entertainment-education through digital storytelling engages learners and enhances discussion and aids understanding of the content.

PrEP4Kink will provide kink-involved participants with an opportunity to receive PrEP information that is culturally tailored to their sexual and community identities, which does not exist in current promotional materials.

PrEP4Kink will measure knowledge of PrEP and attitudes towards PrEP uptake over time. These are elements identified by the Health Belief Model: perceived risk of HIV; susceptibility to HIV; perceived barriers to PrEP uptake; perceived benefits of PrEP uptake; perceived effectiveness of PrEP; and self-efficacy of initiating PrEP uptake. Moderating and ancillary factors will be measured, and their relation to the elements of the Health Belief Model will be analyzed. Moderating factors include the centrality of kink identity; the level of kink community involvement; the types and frequencies of kink and sex behaviors. Demographic variables will be measured and their relation to elements of the Health Belief Model will be analyzed, including age; number of years involved in kink; gender identity; sex assigned at birth; racial/ethnic identity; educational attainment; income level; sexual orientation identity; and sexual attraction.

The primary endpoint is participant-reported uptake of PrEP. This is measured by survey at 3 months, 6 months, 9 months and 12 months of the study. Another primary outcome includes the number of people who persist in using PrEP during the study and the number of pills taken according to clinical guidelines (adherence) since the previous data collection period for each person reporting persistant use of PrEP. These measures will be self-reports at T2 (3 months), T3 (6 months), T4 (9 months) and T5 (12 months) (Please see attachments titled "PrEP4Kink Measures" and "PrEP4Kink Theoretical Framework."

The secondary endpoints are Knowledge about PrEP and Attitudes towards PrEP. The Knowledge about PrEP measure comprises participant-reported items designed to measure key constructs in the Health Belief Model. These participant-reported items will measure perceived benefits of PrEP, the perceived effectiveness of PrEP; perceived risk of HIV acquisition; and perceived susceptibility to HIV acquisition. Items on the survey will also measure perceived barriers to PrEP uptake. Another section of the survey instrument will measure Attitudes towards PrEP. This section will comprise items to measure self-efficacy of initiating PrEP treatment. Another set of items will measure PrEP stigma, including shame, character judgment, and perceived level of social support. Please see attachments titled "PrEP4Kink Measures" and "PrEP4Kink Theoretical Framework."

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Successful completion of screening checklist to indicate one of the following conditions:

  o currently engaging, or have engaged in the last 3 months, in consensual kink activities such as power exchange (Dominant/submissive roles), bondage, sadomasochism, or fetish activities. By fetish, we mean a type of sexual desire in which gratification depends on or is significantly increased by particular objects, clothing items, parts of the body, or types of persons.
* Successful completion of screening checklist to indicate the following conditions:

  * weigh at least 35 kg;
  * report negative HIV serostatus, OR report that they "don't know" their HIV serostatus;
  * has never taken PrEP or been involved in any investigation trial of PrEP medication
* Age of majority in the legal jurisdiction (geographic location) where the survey is taken (usually age 18)
* English-language proficiency sufficient to understand the study instruments
* Completion of an electronically signed and dated informed consent form

Exclusion Criteria:

Individuals will be ineligible for participation if they:

* Are younger than 18 years of age
* Weigh less than 35 kg
* Are currently on PrEP
* Enrolled in an investigational trial of PrEP medication
* Have a self-reported positive HIV serostatus
* Have previously used PrEP but was required to discontinue use due to serious side effects or medical contraindications
* Have been diagnosed with renal failure or are dialysis dependent
* Are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
PrEP Uptake | one year
  Number of participants who test HIV-negative and begin using PrEP, divided by the number of participants who test HIV-negative and are provided information on PrEP through the study. This is a dichotomous variable reported as a percentage.

SECONDARY OUTCOMES:
PrEP Adherence | one year
  Self-report number of pills missed in previous 7 days will be measured every 3 months throughout the implementation period.
Percentage of Treatment Persistence | one year
  Number of people who continue to use PrEP at each T measurement during the study after self-report of starting PrEP, divided by the number of people who use PrEP at previous T measurement (reported as a percentage).

OTHER OUTCOMES:
Knowledge of PrEP | one year
  9 item questionnaire, not a scale
difficulty in initiating PrEP uptake | one year
  self-efficacy of initiating PrEP uptake; 8 item questionnaire, not a scale
Susceptibility to HIV | one year
  3 item modeled on Champion's Health Belief Model Scale, not a scale in this study
Perceived barriers to PrEP uptake | one year
  9 item questionnaire, not a scale
Perceived benefits and effectiveness of PrEP uptake | one year
  3 item questionnaire, not a scale

CONTACTS AND LOCATIONS:
Locations (1):
- TASHRA, Rio Vista, California, United States

REFERENCES:
- [Background] Bauer, R. Queer BDSM intimacies: Critical consent and pushing boundaries. Palgrave: Houndmills 2014.
- [Background] Bauer, R. Desiring masculinities while desiring to question masculinity? How embodied masculinities are renegotiated in les-bi-trans-queer BDSM practices. Norma, 11: 237-254.
- [Background] Bernstein IH, Keith JB. Reexamination of Eisen, Zellman, and McAlister's Health Belief Model questionnaire. Health Educ Q. 1991 Summer;18(2):207-20. doi: 10.1177/109019819101800206. PMID 2055778
- [Background] Bowleg L, Huang J, Brooks K, Black A, Burkholder G. Triple jeopardy and beyond: multiple minority stress and resilience among black lesbians. J Lesbian Stud. 2003;7(4):87-108. doi: 10.1300/J155v07n04_06. PMID 24831386
- [Background] Cantor JM. Is homosexuality a paraphilia? The evidence for and against. Arch Sex Behav. 2012 Feb;41(1):237-47. doi: 10.1007/s10508-012-9900-3. PMID 22282324
- [Background] Costello, A. B., & Osborne, J. (2005). Best practices in exploratory factor analysis: Four recommendations for getting the most from your analysis. Practical Assessment, Research, And Evaluation, 10(1), 7.
- [Background] Cramer RJ, Johnson KL, Nobles MR, Holley SR, Desmarais SL, Gemberling TM, Wright S, Wilsey CN, Van Dorn RA. Lifetime Suicide-Related Behavior, Violent Victimization, and Behavioral Health Outcomes: Results From a Vulnerable Population Needs Assessment. J Interpers Violence. 2021 Jun;36(11-12):5860-5871. doi: 10.1177/0886260518801941. Epub 2018 Sep 28. PMID 30261811
- [Background] Cyril S, Smith BJ, Possamai-Inesedy A, Renzaho AM. Exploring the role of community engagement in improving the health of disadvantaged populations: a systematic review. Glob Health Action. 2015 Dec 18;8:29842. doi: 10.3402/gha.v8.29842. eCollection 2015. PMID 26689460
- [Background] Dawson SJ, Bannerman BA, Lalumiere ML. Paraphilic Interests: An Examination of Sex Differences in a Nonclinical Sample. Sex Abuse. 2016 Feb;28(1):20-45. doi: 10.1177/1079063214525645. Epub 2014 Mar 14. PMID 24633420
- [Background] Gonzales G, Dedania R, Driscoll R. Health Insurance Coverage and Access to Care Among US-Born and Foreign-Born Sexual Minorities. J Immigr Minor Health. 2019 Jun;21(3):540-548. doi: 10.1007/s10903-018-0774-x. PMID 29946865
- [Background] Hammers, C., & Brown III, A. D. (2004). Towards a feminist-queer alliance: a paradigmatic shift in the research process. Social Epistemology, 18(1), 85-101.
- [Background] Holvoet L, Huys W, Coppens V, Seeuws J, Goethals K, Morrens M. Fifty Shades of Belgian Gray: The Prevalence of BDSM-Related Fantasies and Activities in the General Population. J Sex Med. 2017 Sep;14(9):1152-1159. doi: 10.1016/j.jsxm.2017.07.003. Epub 2017 Aug 7. PMID 28781214
- [Background] Jacobs LA. Health beliefs of first-degree relatives of individuals with colorectal cancer and participation in health maintenance visits: a population-based survey. Cancer Nurs. 2002 Aug;25(4):251-65. doi: 10.1097/00002820-200208000-00001. PMID 12181494
- [Background] Jaffee KD, Shires DA, Stroumsa D. Discrimination and Delayed Health Care Among Transgender Women and Men: Implications for Improving Medical Education and Health Care Delivery. Med Care. 2016 Nov;54(11):1010-1016. doi: 10.1097/MLR.0000000000000583. PMID 27314263
- [Background] Johnson MJ, Nemeth LS. Addressing health disparities of lesbian and bisexual women: a grounded theory study. Womens Health Issues. 2014 Nov-Dec;24(6):635-40. doi: 10.1016/j.whi.2014.08.003. Epub 2014 Oct 5. PMID 25287354
- [Background] Kahn JH. Factor Analysis in Counseling Psychology Research, Training, and Practice: Principles, Advances, and Applications. The Counseling Psychologist. 2006;34(5):684-718. doi:10.1177/0011000006286347
- [Background] Kinsey, AC, Pomeroy, WB, Martin, CE, Gebhard, PH. Sexual behavior in the human female. Philadelphia: W. B. Saunders Company, 1953.
- [Background] Krafft-Ebing, Richard von. Psychopathia sexualis: with especial reference to the antipathic sexual instinct: a medico-forensic study. (Franklin S. Klaf, Trans. 12th ed.). Arcade Publishing, Inc.: New York City 1965.
- [Background] Martinez, K. (2020). Overwhelming whiteness of BDSM: A critical discourse analysis of racialization in BDSM. Sexualities, 0(0), 1-16. https://doi.org/10.1177/1363460720932389
- [Background] Meyer IH. Prejudice, social stress, and mental health in lesbian, gay, and bisexual populations: conceptual issues and research evidence. Psychol Bull. 2003 Sep;129(5):674-697. doi: 10.1037/0033-2909.129.5.674. PMID 12956539
- [Background] McConnell EA, Janulis P, Phillips G 2nd, Truong R, Birkett M. Multiple Minority Stress and LGBT Community Resilience among Sexual Minority Men. Psychol Sex Orientat Gend Divers. 2018 Mar;5(1):1-12. doi: 10.1037/sgd0000265. PMID 29546228
- [Background] Mvududu NH, Sink CA. Factor Analysis in Counseling Research and Practice. Counseling Outcome Research and Evaluation. 2013;4(2):75-98. doi:10.1177/2150137813494766
- [Background] Quinn DM, Chaudoir SR. Living with a concealable stigmatized identity: the impact of anticipated stigma, centrality, salience, and cultural stigma on psychological distress and health. J Pers Soc Psychol. 2009 Oct;97(4):634-51. doi: 10.1037/a0015815. PMID 19785483
- [Background] Rehor JE. Sensual, erotic, and sexual behaviors of women from the "kink" community. Arch Sex Behav. 2015 May;44(4):825-36. doi: 10.1007/s10508-015-0524-2. Epub 2015 Mar 21. PMID 25795531
- [Background] Richters J, de Visser RO, Rissel CE, Grulich AE, Smith AM. Demographic and psychosocial features of participants in bondage and discipline, "sadomasochism" or dominance and submission (BDSM): data from a national survey. J Sex Med. 2008 Jul;5(7):1660-8. doi: 10.1111/j.1743-6109.2008.00795.x. PMID 18331257
- [Background] Ross TP, Ross LT, Rahman A, Cataldo S. The bicycle helmet attitudes scale: using the health belief model to predict helmet use among undergraduates. J Am Coll Health. 2010;59(1):29-36. doi: 10.1080/07448481.2010.483702. PMID 20670926
- [Background] Rossman K, Salamanca P, Macapagal K. A Qualitative Study Examining Young Adults' Experiences of Disclosure and Nondisclosure of LGBTQ Identity to Health Care Providers. J Homosex. 2017;64(10):1390-1410. doi: 10.1080/00918369.2017.1321379. PMID 28459379
- [Background] Ryan, R. Attachment, emotion regulation, and gender role issues in BDSM relationships: An exploratory analysis. MA Thesis, Southern Illinois University, Edwardsville 2018.
- [Background] Seelman KL, Colon-Diaz MJP, LeCroix RH, Xavier-Brier M, Kattari L. Transgender Noninclusive Healthcare and Delaying Care Because of Fear: Connections to General Health and Mental Health Among Transgender Adults. Transgend Health. 2017 Feb 1;2(1):17-28. doi: 10.1089/trgh.2016.0024. eCollection 2017. PMID 28861545
- [Background] Sheff, E, Hammers, C. The privilege of perversities: race, class and education among polyamorists and kinksters. Psychology & Sexuality 2011;2: 198-223. https://doi.org/10.1080/19419899.2010.537674
- [Background] Simula, B. L. (2019). Pleasure, power, and pain: A review of the literature on the experiences of BDSM participants. Sociology Compass, 13(3), e12668.
- [Background] Sprott RA, Randall A, Smith K, Woo L. Rates of Injury and Healthcare Utilization for Kink-Identified Patients. J Sex Med. 2021 Oct;18(10):1721-1734. doi: 10.1016/j.jsxm.2021.08.001. Epub 2021 Sep 2. PMID 34481743
- [Background] Waldura JF, Arora I, Randall AM, Farala JP, Sprott RA. Fifty Shades of Stigma: Exploring the Health Care Experiences of Kink-Oriented Patients. J Sex Med. 2016 Dec;13(12):1918-1929. doi: 10.1016/j.jsxm.2016.09.019. Epub 2016 Oct 27. PMID 28340946
- [Background] Zhang Y, Hedo R, Rivera A, Rull R, Richardson S, Tu XM. Post hoc power analysis: is it an informative and meaningful analysis? Gen Psychiatr. 2019 Aug 8;32(4):e100069. doi: 10.1136/gpsych-2019-100069. eCollection 2019. PMID 31552383